CLINICAL TRIAL: NCT02420119
Title: Does Intravenous Iron Therapy Decrease Serum Phosphorous and Vitamin D Levels in Patients With and Without Chronic Renal Failure?
Brief Title: Does Intravenous Iron Therapy Decrease Serum Phosphorous Levels?
Status: Completed | Type: Observational
Sponsor: Frieda Wolf (Other)
Responsible Party: Sponsor-Investigator, Frieda Wolf, Dr frieda wolf, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Other Study IDs: EMC 59-14
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Chronic Renal Failure
Keywords: Iron Therapy; serum phosphates; vitamin D
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non interventional

SUMMARY:
Intravenous iron therapy is common and effective, with few side effects. Two formulations are used, venofer or iron sucrose and ferrlecit, or ferric gluconate.

The association between intravenous iron use and decrease in serum phosphorus and vitamin D levels, with increased fractional excretion of phosphorus, has been observed with older iron preparations, such as saccharated ferric oxide. However, hypophosphatemia and osteomalacia have been reported with iron carboxymaltose, a newer iron formulation. There is no information in the literature about phosphorus and vitamin D levels after treatment with venofer or ferrlecit. We intend to check phosphorus and vitamin D serum levels in our patients prior to and after treatment with these iron formulations.

DETAILED DESCRIPTION:
Intravenous iron replacement has become quite common in cases where oral iron therapy is insufficient or poorly tolerated. Various intravenous iron preparations have been used in patients on dialysis and with chronic kidney disease for many years, however, these patients have severely reduced glomerular filtration rate and are generally hyperphosphatemic.

Although generally safe, certain iron preparations have been associated with severe phosphorus and calcitriol deficiency, caused by elevation in serum levels of fgf23, a phosphaturic humoral factor derived from osteocytes. Fractional excretion of phosphorus is indeed raised in these patients. In some cases phosphorus deficiency, or high fgf23 levels, are so severe that osteomalacia can result . This phenomenon has been observed with saccharated ferric oxide , a preparation commonly used in Japan, and in iron polymaltose . It has also been observed with iron carboxymaltose , a newer iron preparation, now available in Israel. These reports propose that iron causes elevated fgf23 levels, which in turn decreases phosphorus absorption and inhibits 1α-hydroxylase activity. Patients with deficient vitamin D have greater tendency to develop hypophosphatemia.

This phenomenon of phosphorus deficiency has not been documented in the commonly used preparations of iron sucrose (venofer) and ferric gluconate (ferrlecit). These non-dextran iron preparations have a very low rate of allergic reactions and adverse events. They are used in various cases of iron deficiency anemia with normal renal function, such as patients with Inflammatory bowel disease , diabetics or in people who cannot tolerate oral iron therapy. Moreover, certain oral iron preparations are under investigation at present for their role as phosphorus binders.

The purpose of this study is to measure phosphorus, parathyroid hormone and vitamin D levels in patients prior to and after intravenous iron therapy in patients with iron deficiency anemia with normal and reduced Glomerular Filtration Rate . We hypothesize that iron therapy with ferric gluconate and iron sucrose will induce hypophosphatemia and low levels of 1,25 hydroxide Vit D. We will try to ascertain whether the hypophosphatemia is clinically significant or merely a low laboratory value, and whether patients with vitamin 25 hydroxide -D deficiency have a greater propensity to develop it.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Have an indication for intravenous iron treatment
* Estimated Creatinine clearance at least 30ml/min (patients with lower Estimated Creatinine clearance may not be able to excrete phosphorus)
* Have signed informed consent.

Exclusion Criteria:

* Pregnancy
* Estimated creatinine clearance below 30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in a period of one year we will try to recruit approximately 100 men and women over the age of 18, who have iron deficiency anemia and have been prescribed intravenous iron treatment at the ambulatory treatment unit.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to show a mean difference of 0.16 mmol/L for serum phosphorus before and after treatment, samples from 23 patients were needed . we recruited more patients than were needed to demonstrate this difference.
Groups:
- Self-control Observational Cohort: 48 subjects with iron deficiency anemia, had serum phosphorus levels checked before and after administration of intravenous iron.
Period: Overall Study
Arm/Group | Self-control Observational Cohort
Started | 53
Completed | 48
Not Completed | 5
Not completed — insufficient laboratory data | 5

BASELINE CHARACTERISTICS:
Population: patients with iron deficiency anemia
Groups:
- Patients Receiving Intravenous Iron: patients over the age of 18 with iron deficiency anemia, who were referred for intravenous iron treatment, who gave consent to participate
Arm/Group | Patients Receiving Intravenous Iron
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.83 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 48
serum phosphorus levels [Mean (Standard Deviation); unit: mg/dL] | 3.46 (0.5)
vitamin D levels [Mean (Standard Deviation); unit: nmol/L] — Population: missing information regarding 5 participants
  nmol/L
    number analyzed (Participants) | 43
    (all) | 40.67 (23.4)
eGFR [Mean (Standard Deviation); unit: ml/min] — Population: missing data
  ml/min
    number analyzed (Participants) | 25
    (all) | 113 (44.4)

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Serum Levels of Phosphorus in Patients After Treatment With Intravenous Iron.
Description: serum phosphorus levels were measure at baseline, and after intravenous iron administration
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Self-control Observational Cohort
Number analyzed (Participants) | 48
mg/dL | 3.47 (0.55)

ADVERSE EVENTS:
Time Frame: 3 months, duration of iron treatment
Description: adverse events were as per clinical standard of care, and not connected to study outcome, since the trial's intervention was blood testing.
Arm/Group | Self-control Observational Cohort
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No